CLINICAL TRIAL: NCT05038007
Title: Pain After Thoracoscopic Lung Surgery - the Effect of Intercostal Nerve Blockades With Standard Bupivacaine and Liposomal Bupivacaine - a Randomised Controlled Feasibility Trial
Brief Title: Pain After Lung Cancer Surgery - Comparing Traditional Versus Prolonged Release Nerve Blockades
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jannie Bisgaard Stæhr (Other)
Responsible Party: Sponsor-Investigator, Jannie Bisgaard Stæhr, Principal Investigator, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAUH-VATS-01
Record Dates: First submitted 2021-08-25; First posted 2021-09-08 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain; Lung Cancer; Video Assisted Thoracoscopic Surgery; Blockades Neuromuscular; Anesthesia, Local
MeSH Terms: conditions — Pain, Postoperative; Lung Neoplasms | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Bupivacaine Hydrochloride in perioperative intercostal blockades
  Interventions: Drug: Bupivacaine Hydrochloride
- Intervention (Experimental): Liposomal bupivacaine in perioperative intercostal blockades
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — As prior described
  Other Names: Exparel
  Arms: Intervention
Drug: Bupivacaine Hydrochloride — As prior described
  Other Names: Marcaine
  Arms: Control

SUMMARY:
To investigate the effect of liposomal bupivacaine compared with bupivacaine hydrochloride for intercostal blockades for patients undergoing Video-assisted thoracoscopic surgery.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) is a minimally invasive routine procedure. It's less invasive than thoracotomy but postoperative pain is still a problem.

At Aalborg University Hospital, intercostal blockades with bupivacaine is used as standard pain treatment for patients undergoing VATS. Adding adjuvants to the blockades may prolong the effect.

The aim of this study is to examine if intercostal nerve blockades with liposomal bupivacaine improves postoperative pain management compared to intercostal nerve blockades with bupivacaine hydrochloride.

ELIGIBILITY:
Inclusion Criteria:

* Adults independent of sex with an age of ≥ 18 years
* Patients undergoing VATS as a part of either examination or treatment of lung cancer

Exclusion Criteria:

* Patients who are unable to understand oral and written information.
* Patients with known chronic pain in the thorax which have been persisting for at least six months before the day of surgery.
* Pregnant and nursing women.
* Patients with hypersensitivity / allergy / Intolerance to dexamethasone or bupivacaine.
* Patients receiving a planned preoperative epidural blockade during their stay.
* Patients converted to open surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesic effect | 48 hours
  Time in hours to first postoperative administration of Pro Re Nata (PRN) opioids

SECONDARY OUTCOMES:
Total equipotent opioid dose | 48 hours
  Total equipotent opioid dose in milligrams during the first 48 hours after surgery.
Numerical Rating Scale | 48 hours
  Pain intensity on a Numerical Rating Scale ranging from 0 indicating no pain to 10 indicating worst pain imaginable during the first two postoperative days.
Mobilisation | 48 hours
  Time in hours to full mobilisation defined as walking with or without aids.
Opioids at discharge | Not fixed. On average 4 days and a maximum of 3 months.
  Need for opioids at discharge (yes or no and equipotent dosage)
Patient-reported satisfaction of postoperative pain management assessed by self-made questionnaire in Danish | Measured twice. Once 48 hours after surgery and once at non fixed time(on average 4 days and a maximum of 3 months)
  Patients are asked to fill out a questionnaire rating their general satisfaction with pain management and sufficiency of pain treatment on a scale from 0 to 10. The questionnaire also assess whether the patients had any perceived side effects and how uncomfortable they were on a scale from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Jannie Bisgaard, MD, PhD, Principal Investigator — Aalborg University Hospital, department of Anaesthesiology
Locations (1):
- Aalborg University Hospital, Aalborg, Region of Northern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No